CLINICAL TRIAL: NCT06949384
Title: Status of Self-Esteem Among Medical Students of a Medical College: A Descriptive Cross-Sectional Study
Brief Title: Self-Esteem Status Among Medical Students: A Descriptive Study
Status: Completed | Type: Observational
Sponsor: Kathmandu Medical College and Teaching Hospital (Other)
Responsible Party: Principal Investigator, Prajwol Neupane, Medical Student, Kathmandu Medical College and Teaching Hospital
Other Study IDs: SelfEsteemStudy_KMCTH
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Self-esteem Among Medical Students
Keywords: medical students; mental health; prevalence; self concept; self-esteem
MeSH Terms: conditions — Psychological Well-Being | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — This observational study focuses on the measurement of self-esteem in medical students using the Rosenberg Self-Esteem Scale. There is no intervention or treatment applied, and participants are only assessed for their self-esteem levels based on their demographic information.

SUMMARY:
The goal of this observational study is to assess the status of self-esteem in medical students of a medical college, focusing on different academic years, and various sociodemographic factors. The main questions it aims to answer are:

What is the prevalence of low, normal, and high self-esteem among medical students?

How do sociodemographic factors (age, gender, nationality, scholarship status, religion, academic year, education level of parents, occupation of parents, motivation behind choosing medicine as a career) influence self-esteem in medical students?

Since this is an observational study, there is no formal comparison group. Researchers will explore the variations in self-esteem levels based on sociodemographic characteristics.

Participants will complete a semi-structured questionnaire providing demographic details, such as age, gender, academic year, and parental education/occupation, and answering the Rosenberg Self-Esteem Scale.

DETAILED DESCRIPTION:
Self-esteem is the assessment and experience related to self-value, the insight of self-ability as well as the reception of the whole self. Abraham Maslow involved self-esteem in his "hierarchy of human needs" which he depicted it in two forms - the need for respect from others (in the form of recognition, success, and admiration), and the need for self-respect (in the form of self-love, self-confidence, skill, or aptitude).

Despite being a predictor of high academic achievement and overall happiness, very few studies are done in medical students of Nepal. This study aims to assess the status of self-esteem in medical students and compare the prevalence of low, normal and high self-esteem among medical students of different academic years. For this study, Rosenberg Self-Esteem Scale tool is being used. To obtain the data for the study, convenience sampling technique will be used. Research is conducted among medical students of Kathmandu Medical College and Teaching Hospital, from 20th August to 10th September. The sample size is calculated as 227. The data will be collected via a semi-structured questionnaire in the English language via Google Forms. SPSS version 26.0 will be used to analyse the data.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Medical students from first year to final year studying Bachelor in Medicine and Bachelor in surgery at Kathmandu Medical College and Teaching Hospital
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Student studying Bachelor of Dental Surgery and Paramedical Studies
* Those who do not fill up the form completely
* Those who are interns and already graduated from medical college
* Those who do not give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First year to Fourth year medical student studying at Kathmandu Medical College and Teaching Hospital
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Self-esteem level | October 17, 2023 to September 17, 2023
  The primary outcome measure is the level of self-esteem among medical students at Kathmandu Medical College, as assessed using the Rosenberg Self-Esteem Scale. This will help determine the proportion of students with low, normal, or high self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Kathmandu Medical College and Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) to be shared will include all anonymized data relevant to the study, such as demographic information (age, gender, etc.), clinical outcomes, laboratory values, and any other study-specific variables that may have been collected. The IPD will be anonymized to ensure patient confidentiality and in compliance with ethical standards for data privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available from January 2025 to January 2026. IPD and supporting information will be available beginning 6 months after the publication of results and will be accessible for 2 years.
Access Criteria: Access to the IPD and supporting information will be available to researchers who provide a research plan and have the necessary ethical approvals. Researchers can request access via email request to the corresponding author. The data will be provided in a secure format to ensure confidentiality and appropriate use. Additionally, the journal will provide access to the data as part of the publication process, in line with their data sharing policies, once the study results are published